CLINICAL TRIAL: NCT03645343
Title: The Effect of Functional Treatment Using the Activator Versus the Twin Block on the Temporomandibular Joint and the Mandibular Movements in Skeletal Class II Patients: A Randomized Controlled Clinical Trial
Brief Title: The Effect of Functional Treatment of Patients With Backward Positioned Chins on the Jaw Joint and Movements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-09-2018
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Malocclusion, Angle Class II; Retrognathism; TMJ
MeSH Terms: conditions — Malocclusion, Angle Class II; Retrognathia | interventions — Activator Appliances

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Activator (Active Comparator): Patients will be treated using the Activator appliance for one and a half year
  Interventions: Device: Activator
- Twin Block (Experimental): Patients will be treated using the Twin Block appliance for 18 months on average
  Interventions: Device: Twin Block
- Control (No Intervention): Patients will be monitored until the last assessment times in the other groups. This group will serve as a control group

INTERVENTIONS:
Device: Activator — This appliance is constructed in one piece to guide the position of the mandible on closure
  Other Names: Andresen Appliance
  Arms: Activator
Device: Twin Block — This appliance is constructed in two pieces to guide the position of the mandible on closure
  Other Names: Clark's appliance
  Arms: Twin Block

SUMMARY:
Patients with class II malocclusion and retrognathic mandibles will be treated using functional appliances and asses the remodeling that is expected to occur in the temporomandibular joint (TMJ) using cone-beam computed tomography (CBCT) images and we will register mandibular movements using electronic axiograph ( a specific apparatus used to record jaw movements in three dimensions).

There are three groups :

1. Activator Group
2. Twin block Group
3. Control Group with no treatment.

Patients will be allocated to the three groups randomly.

Data will be collected using three different approaches:

* CBCT images before treatment and 12 months after treatment
* Axiograph registrations before treatment and 12 months after treatment

DETAILED DESCRIPTION:
The main purposes of this project are:

1. to evaluate the remodeling effects that would take place in the bone structures of the temporomandibular joint (TMJ) during functional treatment.
2. to evaluate the possible change that may occur in mandibular movements following functional treatment.
3. to evaluate the possible change in the spatial relationship between centric occlusion (CO) and centric relation (CR) following functional treatment

ELIGIBILITY:
Inclusion Criteria:

Class II malocclusion Skeletal class II with retruded mandibles. Old between 10-13 years Healthy TMJ Horizontal or normal growth pattern

Exclusion Criteria:

Patients who have been treated previously Patients with syndromes or congenital deformities Signs or symptoms of temporomandibular disorders.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Change in Glenoid Fossa Height | T1: at one day before the commencement of treatment; T2: after 12 months of treatment
  Glenoid fossa height: the vertical space between the roof and lowest edge of the fossa.
  This measurement will be done on the 3D software (3D OnDemand) using CBCT images
Change in Glenoid Fossa Width | T1: at one day before the commencement of treatment; T2: after 12 months of treatment
  Glenoid fossa width: the horizontal space between the anterior and posterior wall of the fossa.
  This measurement will be done on the 3D software (3D OnDemand) using CBCT images
Change in Articular Eminence Inclination | T1: at one day before the commencement of treatment; T2: after 12 months of treatment
  Articular Eminence inclination: the angle between a horizontal plane and the posterior slope of the articular eminence. This measurement will be done on the 3D software (3D OnDemand) using CBCT images
Change in Condylar Height | T1: at one day before the commencement of treatment; T2: after 12 months of treatment
  Condylar Height: the vertical height of the head of the condyle. This measurement will be done on the 3D software (3D OnDemand) using CBCT images
Change in Condylar Width | T1: at one day before the commencement of treatment; T2: after 12 months of treatment
  Condylar Width: the horizontal width of the head of the condyle. This measurement will be done on the 3D software (3D OnDemand) using CBCT images
Change in Condylar Length | T1: at one day before the commencement of treatment; T2: after 12 months of treatment
  Condylar Length: the mesio-distal length of the head of the condyle. This measurement will be done on the 3D software (3D OnDemand) using CBCT images
Change in Condylar Circumference | T1: at one day before the commencement of treatment; T2: after 12 months of treatment
  Condyle circumference: the outer circumference of the head of the condyle. This measurement will be done on the 3D software (3D OnDemand) using CBCT images
Change in the Anterior Joint Space | T1: at one day before the commencement of treatment; T2: after 12 months of treatment
  Anterior Joint Space: the space between the anterior edge of condyle and the posterior slope of the articular eminence.
  This measurement will be done on the 3D software (3D OnDemand) using CBCT images
Change in the Superior Joint Space | T1: at one day before the commencement of treatment; T2: after 12 months of treatment
  Superior Joint Space: the space between the superior edge of the condyle and the roof of the fossa.
  This measurement will be done on the 3D software (3D OnDemand) using CBCT images
Change in the Posterior Joint Space | T1: at one day before the commencement of treatment; T2: after 12 months of treatment
  Posterior joint space: the space between the posterior edge of the condyle and the posterior board of the fossa.
  This measurement will be done on the 3D software (3D OnDemand) using CBCT images
Change in Border Mandibular Movements | T1: at one day before the commencement of treatment; T2: after 12 months of treatment
  Border mandibular movements will be measured on the axiograph apparatus (called Arcosdigma(R)).
Change in the Discrepancy between CO and CR | T1: at one day before the commencement of treatment; T2: after 12 months of treatment
  CO-CR discrepancy: we will measure distance between centric relation and centric occlusion in three dimensions (sagittal, coronal and axial ). These measurements will be done by an electronic axiograph (Arcosdigma(R))

CONTACTS AND LOCATIONS:
Overall Officials: Abdulmalek Majanni, DDS MSc, Principal Investigator — PhD Student in Orthodontics, University of Damascus Dental School, Damascus; Mohammad Y Hajeer, DDS MSc PhD, Study Chair — Associate Professor of Orthodontics, University of Damascus Dental School, Damascus, Syria; Issam Khoury, DDS MSc PhD, Study Director — Professor of Oral and Maxillofacial Surgery, University of Damascus Dental School, Damascus, SYRIA
Locations (1):
- Orthodontic Department, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aidar LA, Dominguez GC, Yamashita HK, Abrahao M. Changes in temporomandibular joint disc position and form following Herbst and fixed orthodontic treatment. Angle Orthod. 2010 Sep;80(5):843-52. doi: 10.2319/093009-545.1. PMID 20578854
- [Background] Cacho A, Ono T, Kuboki T, Martin C. Changes in joint space dimension after the correction of Class II division 1 malocclusion. Eur J Orthod. 2015 Oct;37(5):467-73. doi: 10.1093/ejo/cju091. Epub 2015 Jan 6. PMID 25564505
- [Background] Arat ZM, Gokalp H, Erdem D, Erden I. Changes in the TMJ disc-condyle-fossa relationship following functional treatment of skeletal Class II Division 1 malocclusion: a magnetic resonance imaging study. Am J Orthod Dentofacial Orthop. 2001 Mar;119(3):316-9. doi: 10.1067/mod.2001.110245. PMID 11244427
- [Background] Chavan SJ, Bhad WA, Doshi UH. Comparison of temporomandibular joint changes in Twin Block and Bionator appliance therapy: a magnetic resonance imaging study. Prog Orthod. 2014 Oct 1;15(1):57. doi: 10.1186/s40510-014-0057-6. PMID 25329768
- [Background] Cimic S, Badel T, Simunkovic SK, Pavicin IS, Catic A. Centric slide in different Angle's classes of occlusion. Ann Anat. 2016 Jan;203:47-51. doi: 10.1016/j.aanat.2015.09.001. Epub 2015 Sep 30. PMID 26434757
- [Background] Clark WJ. The twin block technique. A functional orthopedic appliance system. Am J Orthod Dentofacial Orthop. 1988 Jan;93(1):1-18. doi: 10.1016/0889-5406(88)90188-6. No abstract available. PMID 3422118
- [Background] Costea CM, Badea ME, Vasilache S, Mesaros M. Effects of CO-CR discrepancy in daily orthodontic treatment planning. Clujul Med. 2016;89(2):279-86. doi: 10.15386/cjmed-538. Epub 2016 Apr 15. PMID 27152081